CLINICAL TRIAL: NCT00910455
Title: Phase I, Double-Blind, Placebo-Controlled, Ascending, Single-Dose, Safety, Tolerability and Pharmacokinetic Study of SRX246 Capsules in Healthy Adult Volunteers
Brief Title: Study of SRX246 Capsules in Healthy Adult Volunteers
Acronym: AVN005
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azevan Pharmaceuticals (Industry)
Responsible Party: Neal G. Simon, Ph.D., CEO, Azevan Pharmaceuticals, Inc.
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: AVN005
Record Dates: First submitted 2009-05-27; First posted 2009-05-29 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: Phase 1; Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — SRX246

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Single oral dose of SRX246 capsule
  Interventions: Drug: SRX246
- Placebo (Placebo Comparator): Single oral dose of placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRX246 — single oral dose of SRX246 capsule
  Arms: Active
Drug: Placebo — Single oral dose of placebo capsule
  Arms: Placebo

SUMMARY:
This is the first study of SRX246 in humans, and is being conducted to begin to establish a safety profile of orally administered SRX246.

DETAILED DESCRIPTION:
This protocol represents the first in human study of SRX246, and is being conducted to begin to establish a safety profile, and collect human tolerability and pharmacokinetic data of orally administered SRX246.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females of non-childbearing potential. Female patients should be either post-menopausal or surgically sterile.
2. Age ≥18 and ≤55 years.
3. Body mass index (BMI) of 18.5 to 34.0 kg/m2, inclusive, and a total body weight of >50kg (110 pounds).
4. In good health as determined by medical history, a baseline physical examination, vital signs, clinical laboratory tests and electrocardiogram (ECG) measurement.
5. Subject is willing and able to sign written informed consent prior to receipt of any study medication or beginning study procedures.
6. Subject is willing and able to follow instructions, comply with the protocol requirements and make all required study visits.

Exclusion Criteria:

1. Pregnant or lactating females, or females of childbearing potential.
2. Subject is positive for HIV, hepatitis B surface antigen or hepatitis C antibody tests at screening.
3. Subject with a positive urine test for drugs of abuse or alcohol at screening or at admission to the clinic on study Day -1.
4. Evidence of any out-of range laboratory value at screening that has not been reviewed, approved and documented as not clinically significant by the Principal Investigator.
5. Subject who has resting supine blood pressure outside of a systolic blood pressure range of 90-140 mmHg or a diastolic blood pressure outside a range of 50-90 mmHg on two consecutive measurements taken up to 10 minutes apart.
6. Subject who has resting supine pulse rate greater than 100 bpm or less than 50 bpm on two consecutive measurements taken up to 10 minutes apart.
7. Subject has taken any alcohol within 48 hours of ANY study-related activities AND cannot abstain from drinking alcohol during the entire duration of the subject's study participation.
8. Subject has used any tobacco products in the past 12 months.
9. A history of significant drug allergy or systemic allergic disease (e.g., urticaria, atopic dermatitis).
10. A general medical or psychological condition or behavior, including current substance dependence or abuse that, in the opinion of the investigator, might not permit the subject to complete the study or sign the informed consent.
11. Any clinically significant abnormality on screening 12-lead ECG (e.g., heart block, conduction disorders, ventricular and/or atrial arrhythmias).
12. Any other condition or clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening that, in the opinion of the Principal Investigator or the Physician Sub-Investigator, would make the subject unsuitable for the study or put them at additional risk.
13. Routine or PRN consumption of medications or herbal supplements that the subject is unable or unwilling to discontinue during the study.
14. Inability to understand or follow study instructions.
15. Treatment with an investigational drug within 30 days preceding the first dose of study medication.
16. Known allergy or hypersensitivity to the investigational study drug/placebo components.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability of SRX246 at single doses ranging between 20 and 360 mg | 24 hours

SECONDARY OUTCOMES:
To assess Pharmacokinetics of SRX246 at single doses ranging between 20 and 360 mg | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Benno G Roesch, MD, Principal Investigator — Advanced Biomedical Research
Locations (1):
- Advanced Biomedical Research, Hackensack, New Jersey, United States